CLINICAL TRIAL: NCT02915614
Title: Effects of Pulmonary Rehabilitation on Skeletal Muscle Morphology and Metabolism in PiMM vs. PiZZ COPD Patients
Brief Title: Effects of Pulmonary Rehabilitation on Skeletal Muscle in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician, Department of Respiratory Medicine, Schön Klinik Berchtesgadener Land
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AAT 2016
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: alpha-1 antitrypsin deficiency; pulmonary rehabilitation; exercise training; skeletal muscle biopsy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PiMM patients (Active Comparator): COPD patients with the Alpha-1 antitrypsin genetic variant "PiMM" (Smoking-related COPD)
  Interventions: Procedure: Pulmonary rehabilitation
- PiZZ patients (Experimental): COPD patients with alpha-1 antitrypsin deficiency (genotype PiZZ)
  Interventions: Procedure: Pulmonary rehabilitation

INTERVENTIONS:
Procedure: Pulmonary rehabilitation — 3-weeks of inpatient pulmonary Rehabilitation including exercise Training (daily endurance and strength Training)

SUMMARY:
In a former study, the investigator observed significant differences in the response to pulmonary rehabilitation between COPD patients with the "normal" genetic variant of alpha-1 antitrypsin (PiMM) and those with a homozygous deficient variant (PiZZ) (Jarosch et al., 2016, DOI: 10.1159/000449509). PiZZ COPD patients showed less improvement in exercise capacity compared to PiMM patients. This latter finding was mirrored by an increase of oxidative myofiber type I proportion - that is important for aerobic exercises in daily life - in PiMM but not PiZZ patients.

Based on this finding of impaired skeletal muscle adaptation, the aim of this study is to compare the effects of pulmonary rehabilitation including exercise training on a) specific enzymes of energy metabolism reflecting the oxidative capacity of the skeletal muscle and b) the analogue gene expression of these oxidative enzymes in a cohort of PiMM and PiZZ COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease
* phenotype PiMM or PiZZ
* written informed consent

Exclusion Criteria:

* any comorbidities that prevent patients from participating in an exercise Training program
* necessity of anticoagulant therapy
* other genetic variants of alpha-1 antitrypsin than PiMM or PiZZ

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Endurance time | 3 weeks
  Will be measured during a constant work rate cycling test

SECONDARY OUTCOMES:
Myofibre type I Distribution | 3 weeks
  Skeletal muscle sample will be taken from the M.vastus lateralis via Bergström muscle biopsy needle
Capillary to fibre ratio | 3 weeks
  Skeletal muscle sample will be taken from the M.vastus lateralis via Bergström muscle biopsy needle
muscle strength | 3 weeks
  strength test in the right knee Extensor and flexor

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof., Principal Investigator — Department of respiratory medicine, Schoen Klinik Berchtesgadener Land
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: Undecided